CLINICAL TRIAL: NCT00819143
Title: Collection of Blood and Bone Marrow Samples From Select Patients With CML to Measure Minimal Residual Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090062; 09-H-0062
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-07-13

CONDITIONS: Leukemia
Keywords: Tissue Procurement; Sample Collection; Chronic Myelogenous Leukemia; Laboratory Research
MeSH Terms: conditions — Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Although allogeneic stem cell transplantation is curative in CML, evidence of the BCR-ABL oncogene at low levels is still found in long-term follow-up of survivors. Such low levels of BCR-ABL post-transplant which do not fulfill criteria for molecular relapse are monitored regularly and considered to be suppressed by the GVL effect. Treatment with donor lymphocyte infusions is only instituted when quantifiable BCR-ABL transcript levels rise steadily, indicative of a true molecular relapse .

Similarly, BCR-ABL is still detectable in the majority of CML patients treated with imatinib who achieve complete cytogenetic response, although the amount of BCR-ABL transcripts seem to decline with longer follow-up. With 5 years follow-up of CML patients at CP who received imatinib, the estimated cumulative best rates of complete hematologic response and complete cytogenetic response were 98 percent and 87 percent, respectively10. For the minority of CP-CML patients who do not respond satisfactorily to imatinib, second-generation tyrosine kinase inhibitors are now the recommended next line of treatment.

A major question facing clinicians is whether imatinib and the other more pharmacologically potent second-generation tyrosine kinase inhibitors;can suppress the CML clone at the leukemic stem cell level as effectively as allogeneic stem cell transplantation. This protocol is designed to scientifically compare the treatment responses of patients who are treated with allogeneic stem cell transplantation with patients who receive imatinib or second generation tyrosine kinase inhibitors.

The primary endpoint of this trial will be the proportion of patients who have detected minimal residual disease (DMRD) in primitive CD34 plus progenitor subpopulations no earlier than 60 days from the onset of their respective treatments.

DETAILED DESCRIPTION:
Although allogeneic stem cell transplantation is curative in CML, evidence of the BCR-ABL oncogene at low levels is still found in long-term follow-up of survivors. Such low levels of BCR-ABL post-transplant, which do not fulfill criteria for molecular relapse are monitored regularly and considered to be suppressed by the GVL effect. Treatment with donor lymphocyte infusions is only instituted when quantifiable BCR-ABL transcript levels rise steadily, indicative of a true molecular relapse."

Similarly, BCR-ABL is still detectable in the majority of CML patients treated with imatinib who achieve complete cytogenetic response, although the amount of BCR-ABL transcripts seem to decline with longer follow-up. With 5 years follow-up of CML patients at CP who received imatinib, the estimated cumulative best rates of complete hematologic response and complete cytogenetic response were 98 percent and 87 percent, respectively 10. For the minority of CP-CML patients who do not respond satisfactorily to imatinib, second-generation tyrosine kinase inhibitors are now the recommended next line of treatment.

A major question facing clinicians is whether imatinib and the other more pharmacologically potent second-generation tyrosine kinase inhibitors can suppress the CML clone at the leukemic stem cell level as effectively as allogeneic stem cell transplantation. This protocol is designed to scientifically compare the treatment responses of patients who are treated with allogeneic stem cell transplantation with patients who receive imatinib or second generation tyrosine kinase inhibitors.

The primary endpoint of this trial will be the proportion of patients who have detected minimal residual disease (DMRD) in primitive CD34 plus progenitor subpopulations no earlier than 60 days from the onset of their respective treatments.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Diagnosed with CML
  2. Age 18 years and older

EXCLUSION CRITERIA:

1. Less than 60 days from onset of CML directed treatment
2. Unable to comprehend the investigational nature of the protocol participation or unable to sign their own consent document.
3. Platelet count less than 50 times 10(9)/L (Bone marrow donors only)
4. Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-12-29; Study Completion 2011-07-13

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Cortes J. Natural history and staging of chronic myelogenous leukemia. Hematol Oncol Clin North Am. 2004 Jun;18(3):569-84, viii. doi: 10.1016/j.hoc.2004.03.011. PMID 15271393
- [Background] Vardiman JW, Harris NL, Brunning RD. The World Health Organization (WHO) classification of the myeloid neoplasms. Blood. 2002 Oct 1;100(7):2292-302. doi: 10.1182/blood-2002-04-1199. PMID 12239137
- [Background] Baccarani M, Saglio G, Goldman J, Hochhaus A, Simonsson B, Appelbaum F, Apperley J, Cervantes F, Cortes J, Deininger M, Gratwohl A, Guilhot F, Horowitz M, Hughes T, Kantarjian H, Larson R, Niederwieser D, Silver R, Hehlmann R; European LeukemiaNet. Evolving concepts in the management of chronic myeloid leukemia: recommendations from an expert panel on behalf of the European LeukemiaNet. Blood. 2006 Sep 15;108(6):1809-20. doi: 10.1182/blood-2006-02-005686. Epub 2006 May 18. PMID 16709930